CLINICAL TRIAL: NCT01159353
Title: A Randomized, Double Blind Study to Assess the Pharmacodynamic and Pharmacokinetic Effects of Insulin Glulisine in Obese Subjects With Type 2 Diabetes After a Standard Meal in Comparison to Insulin Aspart
Brief Title: Pharmacodynamic and Pharmacokinetic Effects of Insulin Glulisine in Obese Subjects With Type 2 Diabetes After a Standard Meal in Comparison to Insulin Aspart
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, Sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: APIDR_C_01160; 2006-005536-24 (EudraCT Number)
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2010-07-16 (Estimated); Status verified 2010-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin glulisine; Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- insulin glulisine + insulin aspart (Experimental): insulin glulisine (1 day) + wash-out (7 days) + insulin aspart (1 day)
  Interventions: Drug: Insulin glulisine; Drug: Insulin aspart
- insulin aspart + insulin glulisine (Experimental): insulin glulisine (1 day) + wash-out (7 days) + insulin aspart (1 day)
  Interventions: Drug: Insulin glulisine; Drug: Insulin aspart

INTERVENTIONS:
Drug: Insulin glulisine — Insulin glulisine 100 U/ml, solution for injection in vial Dose: 0.2 U/Kg Administration: single subcutaneous injection with syringe in the periumbilical abdomen within 2 minutes before the standard meal
  Other Names: Apidra
Drug: Insulin aspart — Insulin aspart: 100 U/mL, solution for injection in vial Dose: 0.2 U/Kg Administration: single subcutaneous injection with syringe in the periumbilical abdomen within 2 minutes before the standard meal
  Other Names: NovoRapid

SUMMARY:
Primary Objective:

* To assess the effect of insulin glulisine on the post-prandial plasma glucose excursion during the first hour after a standard meal in comparison to insulin aspart in obese subjects with type 2 diabetes.

Secondary Objectives:

Pharmacodynamic objectives:

* To assess the effect of insulin glulisine on the postprandial plasma glucose excursion during 6 hours after a standard meal in comparison to insulin aspart.

Pharmacokinetic objective:

* To assess post-prandial plasma insulin excursion after a standard meal, in each treatment groups

Safety objective:

* To assess the safety of insulin glulisine in comparison to insulin aspart

DETAILED DESCRIPTION:
Duration of treatment: two study days separated by a 7-day wash-out period

Duration of observation:

* screening period of 1-2 weeks, >2 study days (with a wash-out period of 7 days between the study days),
* Follow-up visit (within 2 weeks after the end of the study treatment period).

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 diabetes for at least one year
* treated with oral antidiabetic agents (OADs) for at least 6 months
* Baseline C-peptide ≥0.1 nmol/L
* BMI (body mass index) between 30 and 40 kg/m2
* HbA1c (glycosylated hemoglobin) < 8.5%
* signed informed consent

Exclusion Criteria:

* type I diabetes mellitus
* current treatment with insulin
* pregnant and breast-feeding women
* any medication known to influence insulin sensitivity
* current treatment with systemic corticosteroids
* history of acute metabolic complications in the past 3 months
* recurrent severe hypoglycaemia or hypoglycaemic unawareness
* active proliferative diabetic retinopathy and known diabetic gastroparesis
* impaired hepatic function, as shown but not limited to ALT or AST above 2 times the upper limit of normal
* clinically relevant illness such as nephropathy and impaired renal function as shown by clearance < 30 ml/min
* any history or presence of clinically relevant abnormality, medical condition (cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, hematological, neurologic, psychiatric, systemic, ocular or infectious disease; any acute infectious disease or signs of acute illness making implementation of the protocol or interpretation of the results difficult
* hypersensitivity to insulins or insulin analogs

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Area under the plasma glucose concentration curve (AUC) between 0 and 1 hour after insulin injection AUC(0-1h) | At day 1 of each treatment period

SECONDARY OUTCOMES:
Area under the curve of plasma glucose concentration AUC(0-2h) | At day 1 of each treatment period
Area under the curve of plasma glucose concentration AUC(0-4h) | At day 1 of each treatment period
Area under the curve of plasma glucose concentration AUC(0-6h) | At day 1 of each treatment period
Delta plasma glucose at 1h after standard meal | At day 1 of each treatment period
Maximum glucose concentration (GLU max) | At day 1 of each treatment period
Maximum glucose excursion (delta GLU max) | At day 1 of each treatment period
Time to delta GLU max | At day 1 of each treatment period
Time to fraction of total glucose AUC(10%, 20%) | At day 1 of each treatment period
Area under the plasma insulin concentration curve AUC (0-1h) | At day 1 of each treatment period
Area under the plasma insulin concentration curve AUC (0-2h) | At day 1 of each treatment period
Area under the plasma insulin concentration curve AUC (0-4h) | At day 1 of each treatment period
Area under the plasma insulin concentration curve AUC (0-6h) | At day 1 of each treatment period
Maximum insulin concentration (Cmax) | At day 1 of each treatment period
Time to fraction of total insulin AUC (10%, 20%) | At day 1 of each treatment period
Time to Cmax | At day 1 of each treatment period
Hypoglycaemia and adverse events | from randomization to the end of study

CONTACTS AND LOCATIONS:
Locations (1):
- Sanofi-Aventis Administrative Office, Paris, France